CLINICAL TRIAL: NCT04953871
Title: Clinical and Ultrasonographic Enthesitis Assessment Before and After Anti-Tumor Necrosis Factor Treatment in Patients With Spondyloarthritis
Brief Title: Enthesitis Assessment Before and After Anti-Tumor Necrosis Factor Treatment in Spondyloarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gunay ER (Other)
Responsible Party: Sponsor-Investigator, Gunay ER, Medical Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 89403766-604.01.02-147611
Record Dates: First submitted 2021-06-22; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Spondyloarthritis; Enthesitis; Anti-Tumor Necrosis Factor Drugs
MeSH Terms: conditions — Spondylarthritis | interventions — Tumor Necrosis Factor Inhibitors

STUDY DESIGN:
Masking Description: All patients were evaluated by the researcher who had a 10-year experience of musculoskeletal ultrasonography and is blind to clinical evaluation.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Spondyloarthritis (Experimental): Spondyloarthritis patients who was initiated TNF alfa blocker
  Interventions: Drug: TNF Inhibitor

INTERVENTIONS:
Drug: TNF Inhibitor — TNF inhibitors are widely used in patients with spondyloarthritis

SUMMARY:
Biological therapies should be considered in patients with high disease activity despite nonsteroid antiinflammatory drug treatment. The first option among biological therapies is anti-Tumor Necrosis Factor (anti-TNF) drugs. In recent years, anti-TNF treatments have shown that clinical and ultrasonographic enthesitis may improve as well as disease activity, quality of life and acute phase reactants. In this prospective study, we aimed to evaluate the clinical and ultrasonographic evaluation of enthesitis and to determine its response to anti-TNF treatment in patients with SpA.In this prospective study, we aimed to evaluate the clinical and ultrasonographic evaluation of enthesitis and to determine its response to anti-TNF treatment in patients with SpA.

ELIGIBILITY:
Inclusion Criteria:

* Spondyloarthritis patients were diagnosed according to 2009 Assessment of Spondyloarthritis International Society (ASAS) criteria

Exclusion Criteria:

* Severe cardiovascular and respiratory diseases,
* Severe liver and kidney failure,
* Pregnancy and lactation,
* Active infection,
* Malignancy,
* Demyelinating diseases,
* Systemic lupus erythematosus,
* History of knee, elbow, foot and ankle surgery,
* Fluoroquinolone, retinoid and fluoride use,
* Local corticosteroid injection at the examination sites within the six weeks before evaluation
* Peripheral neuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
change from ultrasonographic entesitis score at 3 months | before and 3 months after anti-TNF treatment
  Madrid Sonographic Enthesitis Index was used to screen etheseal sites

SECONDARY OUTCOMES:
Change from disease activity | before and 3 months after anti-TNF treatment
  Bath Ankylosing Spondylitis Disease Activity Index was used
Change from disease activity | before and 3 months after anti-TNF treatment
  Ankylosing Spondylitis Disease Activity Score was used
Change from quality of life | before and 3 months after anti-TNF treatment
  Ankylosing Spondylitis Quality of Life was used
Change from Functionality | before and 3 months after anti-TNF treatment
  Bath Ankylosing Spondylitis Functionality Index was used